CLINICAL TRIAL: NCT06772935
Title: Electroacupuncture Treatment of Peripheral Neuropathy After Taxane Chemotherapy for Breast Cancer
Acronym: CIPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHQU-2025001
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; electroacupuncture; taxanes; SNPs; chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: In this study, subjects and evaluators were separated, and statistical analysis was conducted by a dedicated person who was responsible for the non-contact experimental operation process. However, due to the particularity of acupuncture and moxibustion clinical trials, acupuncture and moxibustion specialists are not blinded in the study. And the subjects, researchers, and clinical doctors are unaware of the allocation of research; Only electroacupuncture technicians and research statistics specialists know about the random allocation situation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electroacupuncture+Routine Nursing Group (Experimental)
  Interventions: Behavioral: Electro-acupuncture
- Fake electroacupuncture + Routine Nursing Group (Placebo Comparator)
  Interventions: Behavioral: Electro-acupuncture

INTERVENTIONS:
Behavioral: Electro-acupuncture — A method of acupuncture that combines acupuncture with a certain frequency of electrical stimulation. Electrical stimulation is a mild level of stimulation intensity that is acceptable to the human body.

SUMMARY:
Electroacupuncture treatment of peripheral neuropathy after taxane chemotherapy for breast cancer

DETAILED DESCRIPTION:
Chemotherapy induced peripheral neuropathy has a significant impact on the integrity of chemotherapy cycle and quality of life of breast cancer patients. The latest research reports indicate that electroacupuncture has a certain therapeutic effect on peripheral neuropathy. In addition, existing studies have confirmed that the peripheral neuropathy of breast cancer induced by taxane is related to genetic factors. This study is based on electroacupuncture treatment of peripheral neuropathy induced by paclitaxel drugs, while screening SNPs related to peripheral neuropathy induced by taxane drugs, and establishing a prognostic model. Eligible patients diagnosed as stage I, II or IIIA breast cancer with peripheral neuropathy for at least 2 weeks were assessed by functional cancer treatment assessment/gynecological oncology group neurotoxicity scale (FACT/GOG-NTX) and the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire CIPN Twenty Item Scale (EORTC QLQ-CIPN20). All items in the above two scales are scored using Likert's 5 and 4 levels. The researchers will temporarily divide the study into two groups, and if necessary, the researchers will add this group. Laboratory personnel are unaware of all clinical and outcome data.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients diagnosed by pathology;

  * EOOG score is 0 or 1;

    * The age range for enrollment is between 18 and 75 years old; ④ Accept chemotherapy regimens based on taxane drugs (alone or in combination);

      ⑤ Previously received taxane chemotherapy for more than 6 months;

      ⑥ According to the National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) 5.0, reporting CIPN symptoms of grade 1 or higher for more than 2 weeks;

      ⑦ Voluntarily participate in this clinical trial and sign the informed consent form;
      * Accept regular follow-up visits; ⑨ There is complete pathological data available.

Exclusion Criteria:

* Non breast cancer patients;

  * Received electroacupuncture treatment within 6 months prior to the start of the study;

    * Patients who experience intolerable toxic side effects during standard dose chemotherapy and terminate the chemotherapy cycle;

      * Prior to enrollment, there was a history of peripheral neuropathy;

        * Unstable heart disease or myocardial infarction within the first 6 months of the study;

          ⑥ Active skin diseases or surface skin ulcers or infections that cannot tolerate electroacupuncture treatment;

          ⑦ Uncontrolled epilepsy patients with uncontrolled seizures;

          ⑧ Merge with other malignant tumor patients;

          ⑨ Pregnancy and lactation period;

          ⑩ Refusal to join clinical trial patients

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients diagnosed with breast cancer. Male patients with breast cancer were excluded.
Enrollment: 162 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group Neurotoxicity Index （FACT/GOG-NTX） | After enrollment, the first assessment of the scale will be conducted, followed by another assessment of the scale at the 4th and 8th week of treatment (7 days per week).
  This scale is mainly used to evaluate chemotherapy induced peripheral neuropathy (CIPN), especially the neurotoxic reactions in gynecological tumor treatment. Through this scale, it is possible to quantify the neurotoxic symptoms that patients experience after receiving chemotherapy, such as sensory abnormalities, motor dysfunction, etc., in order to better monitor and manage the patient's health status.

SECONDARY OUTCOMES:
The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire CIPN-20. | After enrollment, the first assessment of the scale will be conducted, followed by another assessment of the scale at the 4th and 8th week of treatment (7 days per week).
  This scale is used to evaluate the impact of chemotherapy induced peripheral neuropathy (CIPN) on the quality of life of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: Undecided